CLINICAL TRIAL: NCT02844725
Title: A Randomized, Double-Blind, Parallel Group, Placebo-Controlled Stdy to Evaluate the Analgesic Efficacy and Safety of VVZ-149 Injection for Post-operative Pain Following Laparoscopic or Robotic-assisted Laparoscopic Gastrectomy
Brief Title: Evaluate the Analgesic Efficacy and Safety of VVZ-149 Injection for Post-operative Pain Following Gastrectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vivozon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PT-VVZ149-05
Record Dates: First submitted 2016-07-17; First posted 2016-07-26 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Post-Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Water; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- VVZ-149 injection (Experimental): VVZ-149 injections will be mixed with saline, then intravenous infusion for 10hr. The drug product will be administrated with a loading dose of 1.8 mg/kg for 0.5 hour followed by a maintenance dose of 1.3 mg/kg/h for 9.5 hours.
  Interventions: Drug: VVZ-149 injections
- Placebo (Placebo Comparator): Placebo group will receive an water for injection the same volume and period of experimental group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VVZ-149 injections — Colorless, transparent liquid in water for injection
  Other Names: VVZ-149 injection
  Arms: VVZ-149 injection
Drug: Placebo — water for injection
  Other Names: water for injection
  Arms: Placebo

SUMMARY:
The purpose of this phase 2 study is to evaluate the efficacy and safety of an analgesic drug candidate, VVZ-149 Injections. The study is designed as randomized, double-blind, parallel, and placebo-controlled study.

DETAILED DESCRIPTION:
VVZ-149 is a dual antagonist of GlyT2 and 5HT2A. GlyT2 blockage increases inhibitory synaptic transmission by glycine in the spinal cord, resulting in a reduction of pain transmissions to the brain. 5HT2A blockage decreases descending serotonergic facilitatory modulation on pain transmission by the brain and reduces nociceptor activation in peripheral nerves, which are primary sources of pain in post-surgical pain. VVZ-149 has been shown to have comparable efficacy to morphine in well controlled (blind, complete randomization with a positive control) animal studies using rat models of post-operative pain and formalin-induced pain. The PK/PD study in animals indicates that therapeutic plasma concentration in human subjects will be 600-1,900 ng/ml. A clinical Phase 1 study performed in healthy subjects has shown no clinically significant adverse events up to a plasma concentration level of 3,261 ng/ml other than brief symptoms of mild nausea or dizziness, and mild somnolence when the plasma exposure level is more than 2,000 ng/ml.

ELIGIBILITY:
Inclusion Criteria:

1. Patient between the ages of 25 and 70 years old
2. Male patient, in the case of female patient, postmenopausal women, or women physically incapable of childbearing
3. Subject who underwent surgery specially for the clinical study
4. Ability to provide written informed consent prior to any study procedures.
5. Ability to understand study procedures and communicate clearly with the investigator and staff.
6. Subjects with body weight under 100kg and body mass index (BMI) level lower than 35 kg/m2, inclusive

Exclusion Criteria:

< Surgical Factors >

1. Emergency or unplanned surgery.
2. Repeat operation (e.g., previous surgery within 30 days for same condition).
3. Cancer-related condition causing preoperative pain in site of surgery.

   < Subject Characteristics >
4. Women with childbearing potential, Women who are pregnant or breastfeeding.
5. Chronic pain diagnosis (e.g., ongoing pain at baseline with NRS ≥ 4/10).
6. Unstable or poorly controlled psychiatric condition (e.g., untreated PTSD, anxiety, or depression). Subjects who take stable doses (same dose >30 days) of antidepressants and anti-anxiety drugs may be included.
7. Unstable or acute medical condition (e.g., unstable angina, congestive heart failure, renal failure, hepatic failure, AIDS).
8. Subjects who have long PR (>200msec) or prolonged QTc (> 450msec in male, >470msec in female) at Screening

   < Drug, Alcohol, and Pharmacological Considerations >
9. History of alcohol, opiate or other drug abuse or dependence within 12 months prior to Screening .
10. Ongoing or recent (within 30 days prior to surgery) use of steroids, opioids, or antipsychotics.
11. Alcohol consumption within 24 hours of surgery.
12. Use of nonsteroidal anti-inflammatory drugs (NSAIDs) or acetaminophen within 24 hours of surgery.
13. Use of herbal agents or nutraceuticals (i.e., chaparral, comfrey, germander, jin bu huan, kava, pennyroyal, skullcap, St. John's wort, or valerian) within 7 days prior to surgery.

    < Anesthetic and Other Exclusion Considerations >
14. Use of neuraxial or regional anesthesia related to the surgery.
15. Use of ketamine, gabapentin, pregabalin, or lidocaine (>1 mg/kg) intra or peri-operatively, or within 24 hours of surgery.
16. Subject with known allergies to hydromorphone.
17. Subjects who received another investigational drug within 30 days of scheduled surgery

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change of Pain Intensity | prior toPCA, at 1, 2, 4, 6, 8, 10, 24 hours post-dose
  Change of Pain Intensity assessed on the Numerical Rating Scale (NRS) using a 10-point scale up to 24 hours

SECONDARY OUTCOMES:
Difference of Opioid Consumption between Study Groups | 0-2, 2-4, 4-6, 6-8, 8-10, 10-12, 12-14, 14-16, 16-18, 18-20, 20-22, 22-24 hours post-dose
Pain Intensity Difference (PID) using Numerical Pain Rating Scale (NRS, 0-10) up to 24 hours | 1, 2, 4, 6, 8, 10, 24 hours post-dose
Global measurement of patient satisfaction assessed on the questionnarie (0-5 points scale) | 10, 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Seonjun Bae, MD, PhD, Principal Investigator — Yonsei University Health System, Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea